CLINICAL TRIAL: NCT07004608
Title: The Effectiveness Of A Community-based Video-facilitated Parenting Intervention For Child Development Integrated Into Routine Maternal And Child Care Services In India: Study Protocol
Brief Title: A Community-based Video-facilitated Parenting Intervention For Child Development In India.
Status: Completed | Type: Observational
Sponsor: Sangath (Other)
Collaborators: UNICEF (Other)
Responsible Party: Principal Investigator, Reetabrata Roy, Principal Investigator, Sangath
Other Study IDs: RR_2019_58; IND/PCA20231309/SPD20232091 (Other Grant/Funding Number: UNICEF office of Andhra Pradesh, Karnataka and Telangana)
Record Dates: First submitted 2025-05-14; First posted 2025-06-04 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Child Development; Child Nutrition and Early Child Development
Keywords: Early Child Development; System integration; ICDS; Anganwadi Worker; Facilitated Video Viewing; Parenting intervention; Child nutrition; First 1000 days of life

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Aalana Palana — Alan Palana is a facilitated video viewing intervention which promotes responsive and sensitive parenting, early learning opportunities and desired nutritional practices for young children and pregnant women. The content not only describes 'WHAT' behaviours caregiver should adopt, 'HOW' they could include these behaviours in their routines but also 'WHY' a particular behaviour is important for their child's development.

SUMMARY:
Aalana Palan designed, implemented and evaluated an integrated early child development & nutrition intervention promoting nurturing care in the first 1000 days of life in Telangana, India. It was developed in collaboration with UNICEF and the Department of Women Development and Child Welfare Telangana.

Aalana Palana in Telugu - implies a caring and nurturing environment provided by caregivers to their children. It promotes an inclusive environment for adequate nutrition, responsive and sensitive caregiving including opportunities for learning. Aalana Palana draws from the Nurturing Care Framework that provides guidance on giving children the best start in their lives.

Aalana Palana was developed through extensive community engagement, using culturally relevant and locally adaptable video content. This participatory approach ensured its acceptability and contributed to its success in addressing critical gaps in child growth and development. It was delivered entirely within the existing Integrated Child Development Scheme which ensured its sustainability. The innovative use of facilitated video-viewing allowed for standardized delivery of evidence-based practices, around optimal nutrition and parenting during the first 1000 days, reducing the burden on frontline workers while improving caregiver engagement and comprehension.

This intervention was used by Anganwadi workers to conduct group and individual counselling sessions with caregivers in their communities. Aalana Palana implemented a transition from traditional paper-based counselling sessions to a video-based, discussion and demonstration led counselling model. Age specific videos promoted responsive and sensitive parenting, early learning opportunities for children & include desired nutritional practices for young children & pregnant women. The content not only describes 'WHAT' behaviours caregiver should adopt, 'HOW' they could include these behaviours in their routines but also 'WHY' a particular behaviour is important for their child's development.

A key strength of this study is its policy relevance. Aalana Palana has been incorporated into the ICDS guidelines for Supplementary Nutrition Program in Telangana, providing a blueprint for scaling similar programs across the country and in other LMICs.

DETAILED DESCRIPTION:
Children thrive developmentally when they are surrounded by systems and relationships that consistently provide nurturing care. This care must operate across both proximal environments, such as the family and community-based workers (CBWs), and distal influences such as supportive social policies, institutional services, and cultural norms. A nurturing home environment includes a sensitivity and responsiveness to a child's health and nutritional needs, regular, developmentally appropriate opportunities for learning, emotionally enriching caregiver interactions, and protection from environmental and psychosocial adversity. These elements are especially vital during the first 1000 days of life, a critical window for brain development for future cognitive, social, and emotional functioning.

While global progress has been made in reducing developmental risk, evidenced by a decline in the number of children under five at risk of not reaching their developmental potential from 279.1 million to 249.4 million between 2004 and 2010, the burden remains high, particularly in South Asia. This is due to social and structural inequities that limit caregivers' access to knowledge, stimulation resources, and health-promoting environments.

Intervention research from LMICs has demonstrated that programs integrating nutrition with responsive caregiving and play activities delivered in the early years, yield significantly better developmental and nutritional outcomes than stand-alone nutritional approaches. Parenting programs that emphasize emotionally attuned and developmentally supportive interactions between caregivers and children are especially effective in improving child cognition, caregiver knowledge, parenting behaviors, and the quality of parent-child engagement. These findings necessitate scaling up parenting interventions as a key strategy to support child development.

However, the practical implementation of such programs at scale faces barriers such as substandard and overburdened health systems in LMICs. CBWs-who serve as the primary bridge between health systems and communities-are tasked with delivering a wide range of services without sufficient training, resources, or institutional support. This can compromise their effectiveness and increase burnout and attrition.

To overcome these limitations, experts advocate for contextually appropriate, scalable delivery mechanisms that leverage and strengthen existing systems. This includes equipping CBWs with tailored training, structured supervision, technological tools, and incentives that suit their work. As key intermediaries, CBWs are uniquely positioned to foster behaviour change within households and communities, provided they are adequately supported.

One promising avenue for such scalable innovation is the use of mobile health technologies, including video-based interventions. These platforms can reduce the cognitive and logistical burden on CBWs by standardizing messaging, providing engaging and repeatable content, and supporting fidelity in delivery. Videos are particularly effective at capturing caregiver attention, illustrating practical skills, and enhancing learning through modelling and storytelling, factors that make them well-suited for low-literacy or resource-constrained environments.

Video-based parenting programs have the potential to enhance early stimulation, improve ECD knowledge among caregivers, increase household safety practices, and promote father engagement. Furthermore, video-viewing combined with facilitated discussion is both feasible and impactful in resource-limited settings, enabling large-scale access to high-quality parenting support. Video-based interventions have been used in LMICs to promote maternal and child nutrition , ECD knowledge, early stimulation, fathers' engagement, household environment safety, child cognition and maternal knowledge of child development.

Study Setting The intervention would be embedded within the ICDS in 30 Anganwadi Centres (AWCs) of three ICDS projects viz., Maheshwaram, Khairtabad, and Alwal in Telangana. AWCs are community creches serving a population of 5000 in urban and 1000 in rural areas and are managed by CBWs called Anganwadi workers (AWWs).

Telangana is the youngest state in India, founded in the year 2014. According to the National Family Health Survey-5 (NFHS-5, 2019-21), child feeding practice indicators in the state were concerning, with only 37.1% children under three months breastfed within one hour of birth, 68.2% children under six months exclusively breastfed, 51.3% children aged 6-8 months receiving solid or semi-solid food along with breast milk and a meagre 9.2% children aged 6-23 months receiving an adequate diet. Also, there was a marked worsening of Under 5 (U5) child anthropometry indicators between NFHS-4 and 5, where U5 stunting went up from 28% to 33.1%, U5 underweight from 28.4% to 31.8%, and U5 wasting from 18.1% to 21.7%. The other key consideration to implement Aalana Palana in Telangana was high mobile ownership in the state, with 96% urban and 91% rural households having a mobile phone, and 60% of women having access to a phone they use themselves.

Development of video content Information synthesis: A desk review of published global research on parenting interventions specifically in LMICs, the Nurturing Care Framework, the WHO Care for Development Package, and the early years learning framework. Resources in the Indian context, such as the Mother and Child Protection card, Home-Based Care for Young Child program guidelines, Poshan Abhiyan, and Intintiki Anganwadi, were also reviewed for content and implementation guidelines.

Blueprint: A blueprint was developed based on this review, findings from Aalana Palana's formative research, multiple consultations with system-level stakeholders, and available resources for content development. Eleven videos were prioritized for development including one video for pregnancy, eight videos for caregivers of children up to two years of age (each video specifically targeting 3-month periods viz., 0-3 months, 4-6 months, 7-9 months, up to 22-24 months), one video for caregivers of children aged 2-5 years and one specifically addressing fathers' involvement in parenting. ECD messages and parent-child interaction activities to be included in each video were listed to build a cohesive narrative for a specific age group, keeping in mind counselling sessions that would be conducted by AWWs and also to prevent information overload.

Scripting: This blueprint guided the iterative development of scripts, initially drafted in English, then translated into Telugu and Hindi. Each English script was reviewed by senior Aalana Palana investigators and representatives from ICDS and UNICEF. Finalized scripts were translated using simple, colloquial, and culturally relevant language. Scripts included learning objectives, visuals, narration, and discussion points.

Video content development: A creative team from Telangana handled pre-production, shooting, and post-production. Videos were filmed in local communities, with AWCs assisting in identifying and selecting pregnant women and caregivers based on Aalana Palana team briefings. Informed consent was obtained from all families before filming.

Families were familiarized with the creative team and equipment to ensure natural, real-life visuals. Daily routines were discussed to schedule shoots at convenient times for capturing key interactions. Caregivers received reference videos and coaching for play activities. Efforts were made to include families of both male and female children from diverse social and religious backgrounds to ensure equitable representation Content and structure of Aalana Palana Videos The videos promote responsive parenting, early learning, and recommended nutritional practices for young children and pregnant women. They explain what behaviours to adopt, how to integrate them into routines, and why they matter for child development.

Each 5-6-minute video is divided into three segments, each focusing on specific parenting practices. Instructions to pause and discuss key points encourage two-way communication between AWWs and viewers, allowing space for questions and reflections. A well-known Telangana-based narrator (sutradhaar) concludes each video with key takeaways and actionable steps. Shorter 1-2-minute versions were also created from the main videos to reinforce specific behaviours and shared directly with caregivers.

Feedback on video content: During the production and post-production phases of the video content development, stakeholders from ICDS, UNICEF and the Sangath team iteratively provided feedback to the creative team. These recommendations on organization of visuals in each video, language used in scripts, voice modulation, and cultural diversity of content were used to refine the videos.

Implementation of Aalana Palana Training plan: In consultation with ICDS and UNICEF, a capacity-building plan was developed and integrated into AWWs' existing training schedules. A three-day, four-hour-per-day training was conducted, emphasizing experiential learning and role plays. Content included session plans, learning objectives, and required competencies for delivering Aalana Palana. Topics covered included the importance of early childhood, responsive caregiving, Aalana Palana's goals and content, two-way communication, delivery processes, and supportive supervision. Videos were uploaded onto AWWs' phones via external drives, and they were trained to select age-appropriate videos for sessions.

In December 2021, 30 AWWs from three ICDS projects, along with their supervisors and Child Development Project Officers, underwent in-person training. Pre and post-tests were done at the beginning and end of each training day to understand any changes in knowledge and obtain feedback about sessions from AWWs.

Session delivery: Qualitative research conducted during the formative stage of Aalana Palana highlighted challenges on time use and workload of AWWs. One of the mitigation strategies that emerged during further consultations with AWWs which could facilitate effective implementation of Aalana Palana was the prioritisation of group over individual counselling sessions. Evidence also indicated benefits of parenting interventions involving group-based sessions on child outcomes, particularly in LMICs. Based on this, AWWs were encouraged to use the Aalana Palana videos primarily during group-based counselling sessions. AWWs started delivering Aalana Palana sessions from January, 2022.

Supportive supervision: The Aalana Palana team conducted at least one in-person supervision visit per month for all 30 AWWs and used a semi-structured questionnaire to observe the sessions. To record session delivery, stickers were placed next to the names of caregivers in existing registers maintained by AWWs.

Building on global evidence and contextual relevance, this protocol outlines a study to implement and evaluate Aalana Palana, a culturally adapted, video-facilitated parenting intervention for caregivers of young children in Telangana, India. The intervention is designed to promote responsive caregiving practices and optimal nutrition in the early years of life. Aalana Palana will be integrated within the existing framework of the ICDS and delivered by frontline community-based workers, specifically trained AWWs. By embedding the intervention within routine maternal and child care services and utilizing pre-loaded video content as the primary delivery modality, the program aims to enhance fidelity, reduce provider burden, and improve caregiver engagement. This study will assess the effectiveness of the intervention in improving child developmental outcomes and the home caregiving environment, and will examine its feasibility as a scalable, low-cost solution for low-resource settings.

ELIGIBILITY:
Inclusion Criteria:

* Primary caregiver of a child aged between 0-3 years
* Resident of the intervention area and likely to remain for the study duration
* Able and willing to provide informed consent

Exclusion Criteria:

* Caregivers of children with severe medical conditions requiring intensive hospital-based care
* Families already enrolled in another similar ECD intervention trial
* Caregivers who do not speak the local language

Ages: 0 Years to 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study population will comprise all primary caregivers of children under 3 years of age residing in the catchment areas of 30 Anganwadi Centres (AWCs) where the Aalana Palana intervention will be implemented.
  A household-level mapping exercise will be conducted within the selected AWC catchment areas to identify eligible caregivers. All eligible participants will be approached for consent to participate in the study. Those who provide informed consent will be enrolled and subsequently classified into two groups based on their self-reported exposure to the intervention:
  Exposed group: Participants who report having seen at least one Aalana Palana video in the three months preceding data collection.
  Unexposed group: Participants who report not having seen any Aalana Palana videos in the same period.
  A three-month reference period will be used to minimise recall bias regarding exposure to the video-based intervention.
Sampling Method: Non-Probability Sample
Enrollment: 1824 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Caregiver Reported Early Development Instruments (CREDI) | From July 2023 to January 2024
  A caregiver-reported population-level measure of early childhood development for children aged 0-36 months, was used to assess child development through easily observable milestones and behaviours, focusing on developmental progress. The tool consists of four domains - motor, language, cognitive and socio-emotional. We used the long-form which comprises 108 items. With permission from the publishers, the Sangath team translated the CREDI in Telugu for use in ASPIRE. The Telugu version of the form can be found on their website.

SECONDARY OUTCOMES:
The Family Care Indicators (FCI) questionnaire | From July 2023 to January 2024
  Developed by UNICEF, is a caregiver report used to measure the home environment. Adapted from the Home Observation for Measurement of the Environment (HOME) inventory, it focuses on caregiving practices that support early child development in children aged 0-5 years, particularly in LMICs. The FCI uses yes/no questions to evaluate sources of play materials, variety of play materials, and play activities
The Infant and Young Child Feeding (IYCF) framework | From July 2023 to January 2024
  Used to evaluate child nutrition by collecting data on feeding practices critical for growth and development in children under two years, focusing on breastfeeding and complementary feeding adequacy. It includes a total of 17 indicators recommended by the WHO and UNICEF with operational definitions to measure each indicator. In this study we used the composite indicator of Minimum Acceptable Diet (MAD) which is defined as the percentage of children 6-23 months of age who consumed a minimum acceptable diet during the previous day.

CONTACTS AND LOCATIONS:
Overall Officials: Gauri Divan, Principal Investigator — Sangath
Locations (1):
- Sangath, Goa, India

IPD SHARING:
Plan to Share IPD: Yes
The complete raw dataset, accompanied by a detailed data dictionary explaining each variable and the study's analysis plan, will be made available to interested researchers. Data access will begin one year after publication and remain open indefinitely. Individuals or institutions wishing to use the data may submit a request by contacting the corresponding author via email. Access will be provided upon approval and, if required, the signing of a data access agreement with the senior investigators of the program. This approach aims to promote transparency, encourage secondary analyses, and support collaborative research efforts in the field.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Beginning 1 year after publication with no end date

REFERENCES:
- [Background] Nelson AK, Griest CJ, Munoz LM, Rumaldo N, Miller AC, Soplapuco GM, Lecca L, Shin SS, Acuna LR, Valdivia YV, Ramos AR, Ahumada DG, Ramos BRH, Mejia SA, Serrano EO, Castro WH, Oliva VE, Heyman AS, Hartwell LP, Blackwell RL, Diaz DF, Vibbert MM. Proof of concept of the Universal Baby video innovation for early child development in Lima, Peru. J Pediatr Psychol. 2025 Jan 1;50(1):51-62. doi: 10.1093/jpepsy/jsae035. PMID 38872286
- [Background] Antelman G, Ferla J, Gill MM, Hoffman HJ, Komba T, Abubakar A, Remes P, Jahanpour O, Mariki M, Mang'enya MA, van de Ven R. Effectiveness of an integrated multilevel early child development intervention on caregiver knowledge and behavior: a quasi-experimental evaluation of the Malezi program in Tanzania. BMC Public Health. 2023 Jan 4;23(1):19. doi: 10.1186/s12889-022-14956-2. PMID 36600280
- [Background] Feil EG, Baggett K, Davis B, Landry S, Sheeber L, Leve C, Johnson U. Randomized control trial of an internet-based parenting intervention for mothers of infants. Early Child Res Q. 2020 1st Quarter;50(Pt 1):36-44. doi: 10.1016/j.ecresq.2018.11.003. Epub 2018 Dec 8. PMID 32863565
- [Background] Webster-Stratton C, Kolpacoff M, Hollinsworth T. Self-administered videotape therapy for families with conduct-problem children: comparison with two cost-effective treatments and a control group. J Consult Clin Psychol. 1988 Aug;56(4):558-66. doi: 10.1037//0022-006x.56.4.558. No abstract available. PMID 3143750
- [Background] Feroz A, Jabeen R, Saleem S. Using mobile phones to improve community health workers performance in low-and-middle-income countries. BMC Public Health. 2020 Jan 13;20(1):49. doi: 10.1186/s12889-020-8173-3. PMID 31931773
- [Background] Winters N, Langer L, Geniets A. Scoping review assessing the evidence used to support the adoption of mobile health (mHealth) technologies for the education and training of community health workers (CHWs) in low-income and middle-income countries. BMJ Open. 2018 Jul 30;8(7):e019827. doi: 10.1136/bmjopen-2017-019827. PMID 30061430
- [Background] Scott K, Beckham SW, Gross M, Pariyo G, Rao KD, Cometto G, Perry HB. What do we know about community-based health worker programs? A systematic review of existing reviews on community health workers. Hum Resour Health. 2018 Aug 16;16(1):39. doi: 10.1186/s12960-018-0304-x. PMID 30115074
- [Background] Jaskiewicz W, Tulenko K. Increasing community health worker productivity and effectiveness: a review of the influence of the work environment. Hum Resour Health. 2012 Sep 27;10:38. doi: 10.1186/1478-4491-10-38. PMID 23017131
- [Background] Grantham-McGregor SM, Walker SP. Early Childhood Interventions: Issues to Consider in Getting to Scale. Pediatrics. 2023 May 1;151(Suppl 2):e2023060221P. doi: 10.1542/peds.2023-060221P. No abstract available. PMID 37125888
- [Background] Jeong J, Franchett EE, Ramos de Oliveira CV, Rehmani K, Yousafzai AK. Parenting interventions to promote early child development in the first three years of life: A global systematic review and meta-analysis. PLoS Med. 2021 May 10;18(5):e1003602. doi: 10.1371/journal.pmed.1003602. eCollection 2021 May. PMID 33970913
- [Background] Dulal S, Prost A, Karki S, Saville N, Merom D. Characteristics and effects of integrated nutrition and stimulation interventions to improve the nutritional status and development of children under 5 years of age: a systematic review and meta-analysis. BMJ Glob Health. 2021 Jul;6(7):e003872. doi: 10.1136/bmjgh-2020-003872. PMID 34321232
- [Background] Black MM, Walker SP, Fernald LCH, Andersen CT, DiGirolamo AM, Lu C, McCoy DC, Fink G, Shawar YR, Shiffman J, Devercelli AE, Wodon QT, Vargas-Baron E, Grantham-McGregor S; Lancet Early Childhood Development Series Steering Committee. Early childhood development coming of age: science through the life course. Lancet. 2017 Jan 7;389(10064):77-90. doi: 10.1016/S0140-6736(16)31389-7. Epub 2016 Oct 4. PMID 27717614

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-05-14): https://cdn.clinicaltrials.gov/large-docs/08/NCT07004608/Prot_SAP_000.pdf
  • Informed Consent Form (2023-01-03): https://cdn.clinicaltrials.gov/large-docs/08/NCT07004608/ICF_001.pdf